CLINICAL TRIAL: NCT04183673
Title: Efficacy of Laser + Cryo-thermal Therapy in Rehabilitation Following Total Knee Replacement Surgery: a Randomized Controlled Trial
Brief Title: Laser + Cryo-thermal Therapy Following Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2200 CE
Record Dates: First submitted 2019-11-19; First posted 2019-12-03 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Knee Arthropathy
Keywords: Laser Therapy; Cryotherapy; Thermotherapy; Rehabilitation; knee replacement
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-cryo-usual care (Experimental): Sessions 5 days a week for 3 weeks. Each session includes laser therapy+ cryo-thermal followed by standard rehabilitation program
  Interventions: Procedure: Laser therapy-cryo thermal therapy
- usual care (Active Comparator): Sessions 5 days a week for 3 weeks. Each session includes only standard rehabilitation program
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Laser therapy-cryo thermal therapy — 5 days per week, 3 weeks, sessions including laser therapy + cryo therapy followed by usual rehabilitation
  Arms: Laser-cryo-usual care
Procedure: Usual care — 5 days per week, 3 weeks, sessions of usual rehabilitation
  Arms: usual care

SUMMARY:
Objective To investigate the effectiveness of the use of the QMD Helios Laser device in association with standard rehabilitation therapy in reducing inflammatory symptoms in patients following total knee replacement.

Design Randomized controlled trial. Setting Rehabilitation structure, inpatient Main outcome measures Pain subscale of the WOMAC and Lequesne's Algo-Functional Index (LIKERT scale), knee circumference (measured at the middle line of the knee joint space) and knee flexion /extension range of motion by goniometer.

DETAILED DESCRIPTION:
As life expectancy increases, more and more people are afflicted with degenerative joint diseases. Knee osteoarthritis is a pathology typical of old age (over 60 years), but it can also occur in younger people (aged 40-50 years) and is more prevalent in women (11%) than men (7%). Total knee replacement surgery is becoming increasingly frequent.In the immediate post-operative period, the main problems encountered by patients are: inflammation, edema and, above all, pain. These can strongly influence the restoring of a correct muscle-joint function and hence the time needed for a return to normal activities of daily living (ADLs).Post-operative rehabilitation is now a fundamental part of the functional recovery of patients after knee replacement surgery. Traditional rehabilitation programs are mainly focused on improving joint mobility, reducing musculotendinous retractions, increasing muscle strength and establishing a correct gait pattern. Over the years, in addition to the manual rehabilitative techniques, the use of instrumental methods to stimulate the healing processes and speed up recovery times has become a frequent practice, especially for the management of post-operative pain and inflammation. One of these methods is laser therapy, which consists of light radiation composed of a beam of photons with specific physical characteristics that interacts with living tissue to produce an anti-inflammatory, analgesic and biostimulation effect. Another form of instrumental therapy used in rehabilitation for the management of pain/edema resulting from an inflammatory process is the application of cold (cryotherapy) or heat (thermotherapy) or both together in combination (contrast therapy). Cryotherapy is a type of physical therapy that produces temporary anesthesia of the part undergoing treatment.Thermotherapy consists of the application of heat to stimulate a biological process inducing the release of chemotactic substances and growth factors, which have a powerful regenerative and reparative action. An innovative device that combines the therapeutic advantages of these different forms of physical therapy is QMD Helios (Hakomed, Egna, BZ, Italy), designed to provide cryo-thermal and laser treatment. The device is equipped with a high-power diode laser. This therapeutic laser can work at 3 different wavelengths (808 nm,1064 nm, 1120 nm). The wavelengths are each individually controlled and can be delivered in various modes: continuous wave, pulsed mode, super pulse, and Harmonic pulsation (laser wave emission with a variable frequency - determined by means of a scan performed by the device - suited to the tissue to be treated). This innovative triple-wavelength emission represents the most versatile solution when one wishes to obtain different therapeutic effects at the same time. In addition to the use of laser, the device allows the application of cryo-thermal therapy, simultaneously or separately. Simultaneous administration promotes thermal shock, a basic principle of contrast therapy characterized by a marked variation of temperature (30-40 degrees) within a short space of time (30-60 seconds) inducing vasodilation through the heat and vasoconstriction through the cold. Thermal shock is effective in the early stages of rehabilitation for a rapid resolution of pain and swelling.Although in recent years instrumental therapy has come to play a very important role in rehabilitation medicine in the management of pain/inflammation in the acute patient, there is lack of reported evidence in the literature on the use of laser therapy in patients after knee replacement surgery. The aim of this study is to evaluate the effectiveness of the use of the QMD Helios laser device in association with standard rehabilitation therapy in reducing edema and pain symptoms in patients following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* good general physical conditions
* first total knee replacement

Exclusion Criteria:

* diabetic neuropathy
* renal or hearth disease
* allergic reactions
* Reynaud's disease
* lupus
* rheumatoids arthritis
* peripheral vascular disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Womac Pain subscale | Before treatment (admission) and after treatment (3 weeks after admission)
  Pain subscale of the Western Ontario and McMaster Universities Activity Index (scored on a five point (0-4) LIKERT scale)
Change in knee circumference | Before treatment (admission) and after treatment (3 weeks after admission)
  Knee circumference measured at the middle line of the knee joint space
Change in Lequesne's algo Functional Index | Before treatment (admission) and after treatment (3 weeks after admission)
  Lequesne's algo Functional Index (scored on a five point (0-4) LIKERT scale)

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri, Montescano Rehabilitation Center, Montescano, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No